CLINICAL TRIAL: NCT04037098
Title: Efficiency and Safety of Magnesium Lactate Administration in the Reduction of Gestational Diabetes Incidence.
Brief Title: Magnesium Lactate in the Reduction of Gestational Diabetes Incidence.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of financial support and pandemia
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Fernando Guerrero Romero MD, Head of the research unit, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R-2019-785-040
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Intervention Model Description: Study groups:
  Intervention group. Women 19 to 35 years of age, in the twelfth week of pregnancy, who will receive magnesium lactate, 2 tablets orally every 12 hours (equivalent to 360 mg of elemental magnesium) for 3 months plus baseline dietary magnesium requirement.
  Control group. Women 19 to 35 years of age, in the twelfth week of pregnancy, who will receive 2 tablets orally every 12 hours of on inert placebo for three months plus baseline dietary magnesium requirement.
Who Masked: Participant, Care Provider
Masking Description: Neither the patient nor the treating doctor will know the study group the participant was randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium (Experimental): Magnesium lactate, 2 tablets orally every 12 hours (equivalent to 360 mg of elemental magnesium) for 3 months plus baseline dietary magnesium requirement.
  Interventions: Dietary Supplement: Magnesium lactate.
- Control (Placebo Comparator): 2 tablets orally every 12 hours of on inert placebo for three months plus baseline dietary magnesium requirement.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium lactate. — 2 tablets orally every 12 hours (equivalent to 360 mg of elemental magnesium) for 3 months
  Arms: Magnesium
Dietary Supplement: Placebo — 2 tablets orally every 12 hours of on inert placebo for three months
  Arms: Control

SUMMARY:
Gestational diabetes, occurs during the second or third trimester of pregnancy, with no prior history of diabetes; this entity can be resolved at the end of pregnancy. Magnesium is the fourth most abundant mineral in the body, It plays an essential role in the regulation of insulin metabolism, in the functions of adenosine triphosphate. In Mexico, the prevalence of hypomagnesemia is 36.3% for women. Findings suggesting that magnesium supplementation may be a beneficial indication in metabolic glucose disorders. The hypothesis of this study is: that Magnesium lactate administration is safe and reduces the incidence of gestational diabetes.

DETAILED DESCRIPTION:
Objective: This study aims to evaluate the efficacy and safety of magnesium lactate oral administration in reducing the gestational diabetes incidence.

Design: Randomized, double-blind, placebo-controlled clinical trial.

Study population: Pregnant women aged 19 to 35 years, in the twelfth week of pregnancy, whit hypomagnesemia and without the concomitant disease.

Study groups: an intervention group and a control group.

Sample size: It was calculated using a statistical power of 80%, an alpha value of 0.05; 15% of the difference in the mean of gestational diabetes incidence control group and intervention groups was considered. The estimated sample size was 110 subjects for each group.

Process: All eligible participants according to inclusion and exclusion criteria, will be randomized to one of the study groups.

The intervention group will receive magnesium lactate, 2 tablets orally every 12 hours (equivalent to 360 mg of elemental magnesium) for 3 months plus baseline dietary magnesium requirement; the control group will receive 2 tablets orally every 12 hours of on inert placebo for three months plus baseline dietary magnesium requirement.

The blood concentrations of glucose, triglycerides, magnesium, creatinine, transaminases, and thyroid hormones will be measured, as well as the anthropometric measurements, at baseline and end conditions. Also, an oral glucose tolerance curve will be realized at the 20th gestation week.

Statistical analysis: Numerical values will be expressed as mean ± standard deviation; categorical variables will be expressed as proportions. Differences between the groups were estimated by unpaired Student t-test for numerical variables (Mann-Whitney U test for skewed data) or Chi-square and Fisher´s exact test for categorical variables. Intragroup differences were estimated by paired Student t-test.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 19 to 35 years.
* 12th to 14th gestation weeks.
* Informed consent of the participant.

Exclusion Criteria:

* Diabetes.
* High blood pressure.
* Hypertriglyceridemia (>250 g/dL)
* Neoplasia disease.
* Thyroid disease.
* Hepatic disease.
* Consumption of alcoholic beverages.
* Smoking.
* Medication use (thiazide diuretics, anti-blocking agents, calcium antagonists, statins, nicotinic acid, phenytoin, valproic acid, antidepressants, beta-adrenergic, theophylline, glucocorticoids, in the last year)

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 0 (Actual)
Dates: Start 2022-07-31 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Decreased of gestational diabetes incidence | Three months.
  The incidence of gestational diabetes will be considered as a decrease, at the small proportion difference of less than 13.4% between the incidence of gestational diabetes in the intervention group and the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando PD Guerrero, Principal Investigator — Instituto Mexicano del Seguro Social; Luis PD Simental, Study Chair — Instituto Mexicano del Seguro Social; Gerardo PD Martínez, Study Chair — Instituto Mexicano del Seguro Social; Cludia PD Gamboa, Study Chair — Instituto Mexicano del Seguro Social
Locations (1):
- Biomedical Research Unit. IMSS. Durango, Durango, Durango, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mack LR, Tomich PG. Gestational Diabetes: Diagnosis, Classification, and Clinical Care. Obstet Gynecol Clin North Am. 2017 Jun;44(2):207-217. doi: 10.1016/j.ogc.2017.02.002. PMID 28499531
- [Background] Kim C. Maternal outcomes and follow-up after gestational diabetes mellitus. Diabet Med. 2014 Mar;31(3):292-301. doi: 10.1111/dme.12382. PMID 24341443
- [Background] Al-Badri MR, Zantout MS, Azar ST. The role of adipokines in gestational diabetes mellitus. Ther Adv Endocrinol Metab. 2015 Jun;6(3):103-8. doi: 10.1177/2042018815577039. PMID 26137214
- [Background] Fan Y, Xu R, Cai L, Cai L. [Risk factors of gestational diabetes mellitus among the re-birth pregnant women in Xiamen City in 2015-2016]. Wei Sheng Yan Jiu. 2017 Nov;46(6):925-929. Chinese. PMID 29903201
- [Background] Sarrafzadegan N, Khosravi-Boroujeni H, Lotfizadeh M, Pourmogaddas A, Salehi-Abargouei A. Magnesium status and the metabolic syndrome: A systematic review and meta-analysis. Nutrition. 2016 Apr;32(4):409-17. doi: 10.1016/j.nut.2015.09.014. Epub 2015 Oct 23. PMID 26919891
- [Background] Asemi Z, Karamali M, Jamilian M, Foroozanfard F, Bahmani F, Heidarzadeh Z, Benisi-Kohansal S, Surkan PJ, Esmaillzadeh A. Retracted: Magnesium supplementation affects metabolic status and pregnancy outcomes in gestational diabetes: a randomized, double-blind, placebo-controlled trial. Am J Clin Nutr. 2015 Jul;102(1):222-9. doi: 10.3945/ajcn.114.098616. Epub 2015 May 27. PMID 26016859 (Retraction: PMID 33966085 Am J Clin Nutr. 2021 May 8;113(5):1383)
- [Background] Han H, Fang X, Wei X, Liu Y, Jin Z, Chen Q, Fan Z, Aaseth J, Hiyoshi A, He J, Cao Y. Dose-response relationship between dietary magnesium intake, serum magnesium concentration and risk of hypertension: a systematic review and meta-analysis of prospective cohort studies. Nutr J. 2017 May 5;16(1):26. doi: 10.1186/s12937-017-0247-4. PMID 28476161
- [Background] Dalton LM, Ni Fhloinn DM, Gaydadzhieva GT, Mazurkiewicz OM, Leeson H, Wright CP. Magnesium in pregnancy. Nutr Rev. 2016 Sep;74(9):549-57. doi: 10.1093/nutrit/nuw018. Epub 2016 Jul 21. PMID 27445320
- [Background] Makrides M, Crosby DD, Bain E, Crowther CA. Magnesium supplementation in pregnancy. Cochrane Database Syst Rev. 2014 Apr 3;2014(4):CD000937. doi: 10.1002/14651858.CD000937.pub2. PMID 24696187
- [Background] Guerrero-Romero F, Rodriguez-Moran M. [Oral magnesium supplementation: an adjuvant alternative to facing the worldwide challenge of type 2 diabetes?]. Cir Cir. 2014 May-Jun;82(3):282-9. Spanish. PMID 25238470
- [Background] Morton A. Hypomagnesaemia and pregnancy. Obstet Med. 2018 Jun;11(2):67-72. doi: 10.1177/1753495X17744478. Epub 2018 Mar 7. PMID 29997688
- [Background] Alves JG, de Araujo CA, Pontes IE, Guimaraes AC, Ray JG. The BRAzil MAGnesium (BRAMAG) trial: a randomized clinical trial of oral magnesium supplementation in pregnancy for the prevention of preterm birth and perinatal and maternal morbidity. BMC Pregnancy Childbirth. 2014 Jul 8;14:222. doi: 10.1186/1471-2393-14-222. PMID 25005784
- [Background] Dainelli L, Prieto-Patron A, Silva-Zolezzi I, Sosa-Rubi SG, Espino Y Sosa S, Reyes-Munoz E, Lopez-Ridaura R, Detzel P. Screening and management of gestational diabetes in Mexico: results from a survey of multilocation, multi-health care institution practitioners. Diabetes Metab Syndr Obes. 2018 Apr 5;11:105-116. doi: 10.2147/DMSO.S160658. eCollection 2018. PMID 29670384
- [Background] Ramirez-Torres MA. The importance of gestational diabetes beyond pregnancy. Nutr Rev. 2013 Oct;71 Suppl 1:S37-41. doi: 10.1111/nure.12070. PMID 24147923